CLINICAL TRIAL: NCT03678610
Title: Latrunculin A and Ionomycin as a Handling Medium for ICSI
Brief Title: Handling Medium for ICSI With Ionomycin and Latrunculin A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Banoon IVF Center (Other); Qena Fertility Center (Unknown)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Ibnsina-ICSI-ionomycin-LA
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Ionomycin; latrunculin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICSI medium supplemented with Ionomycin and Latrunculin A (Experimental)
  Interventions: Other: Doing ICSI I a medium supplemented with Ionomycin and Latrunculin A
- ICSI medium as it is (No Intervention)

INTERVENTIONS:
Other: Doing ICSI I a medium supplemented with Ionomycin and Latrunculin A — Ionomycin and Latrunculin A would activate oocyte during ICSI along with cytoskeleton stabilization for a favourable outcomes
  Arms: ICSI medium supplemented with Ionomycin and Latrunculin A

SUMMARY:
Using Latrunculin A and Ionomycin would improve the outcome of ICSI if the handling medium during the ICSI procedure has them.

ELIGIBILITY:
Inclusion Criteria:

* indication for ICSI

Exclusion Criteria:

-

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 700 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Fertilization rate | 6 days of culture

SECONDARY OUTCOMES:
Rates of Blastocyst formation and quality | 6 days of culture
  Number of formed blastocysts and blastocysts with good-quality per fertilized oocytes
embryo utilization rate | 6 days of culture
clinical pregnancy rate | three months
ongoing pregnancy rate | 12 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Qena Fertility Center, Qina, Qena Governorate
  - Banon Assiut, Asyut
  - IbnSina IVF Center, Sohag

IPD SHARING:
Plan to Share IPD: No